CLINICAL TRIAL: NCT04266353
Title: Mechanisms in IGF2 Induced Chemoresistance and Mitochondrial Regulation in Triple Negative Breast Cancer
Brief Title: Effect of Resveratrol on Serum IGF2 Among African American Women
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Gayathri Nagaraj, Principle Investigator, Loma Linda University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 5160378
Record Dates: First submitted 2020-01-27; First posted 2020-02-12 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Chemoprevention
MeSH Terms: interventions — Resveratrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single arm (Experimental): Participants with receive resveratrol at 150 mg daily for 6 weeks
  Interventions: Dietary Supplement: Resveratrol (RSV)

INTERVENTIONS:
Dietary Supplement: Resveratrol (RSV) — Participants will receive Resveratrol at 150 mg daily for 6 weeks.
  Other Names: ResVida

SUMMARY:
African American (AA) women with breast cancer (BC) have higher mortality and are associated with worse outcomes when treated with available adjuvant treatments. Addressing this survival disparity will depend on identifying contributing biologic factors that can be translated into new treatments. Preclinical studies have shown that Insulin-like growth factor-II (IGF-II)expression was significantly higher in AA cell lines and tissue samples when compared to Caucasians indicating that IGF-II is an important biologic factor contributing to higher breast cancer mortality in AA women and is also responsible for chemoresistance in BC cells. In addition preclinical studies also demonstrated that resveratrol (RSV) inhibits IGF-II and induces apoptosis in BC cell lines. Researchers want to test IGF-II levels at baseline in healthy African American women and monitor levels while on resveratrol therapy for 6 weeks.

DETAILED DESCRIPTION:
Resveratrol (RSV) is a naturally occurring polyphenol found in many plants including grapes, peanuts and berries. Resveratrol has attracted a lot of research attention based on preclinical data showing anti-inflammatory and anti-oxidative properties through several mechanisms.RSV is available as over the counter supplement in the United States. Various formulations and dosage forms have been used in previous studies involving cardiovascular health, metabolism and chemoprevention. ResVida®, is an oral preparation consisting of pure trans-resveratrol with a purity of > 99% manufactured by DSM nutritional products will be used in this study. Healthy African American women will receive 1 capsule daily of 150 mg.

Objectives: To test the effects of resveratrol on IGF-II level in healthy AA women.

Eligibility: Healthy adult African American female (18 years of age or older) Design: The study involves an initial visit and 3 additional visits at 2 week interval. At the initial visit, women will participate in a short-talk session to present the study, facts about breast cancer, RSV and protocol requirements. Participants will be evaluated for meeting basic eligibility criteria by a Breast Oncologist. All interested participants will sign an informed consent form and will be provided with a questionnaire to complete. The Oncologist will obtain medical history, use of medication, supplements etc. from consented participants. Consented participants will then meet with the study coordinator who will assign each participant with a study identification (ID) number along with other basic assessment as noted below. The study coordinator will also dispense a 2 week supply of RSV along with a medication calendar to each participant at their initial visit and at visits 2-4. In addition, the participants will have their blood sample collected by a trained phlebotomist during visit 1 and at visits 2-4. Collected blood vials will be handed to research laboratory to determine IGF2 levels as well as other research biomarkers.

ELIGIBILITY:
INCLUSION CRITERIA

* African American ethnicity self-identified
* Female participants aged 18 years and above
* Able to provide written informed consent and to understand, participate and comply with protocol requirements
* Able to comprehend and complete forms in English
* Able to swallow oral capsules
* Willingness to stop dietary supplements and vitamins for the duration of the study
* No history of cancers in the past 5 years
* Willingness to abstain from ingestion of large quantities of RSV containing foods and less than 3 drinks of wine per week.

EXCLUSION CRITERIA

* Pregnant or planning to be pregnant or breast feeding
* Participating in any other clinical study
* History of Diabetes defined as recent A1C greater than 6.5 and or fasting serum glucose greater than or equal to 126 mg/dl
* Self-reported history of major organ dysfunction (renal dysfunction described as glomerular filtration rate (GFR) less than 60 ml/min, liver function tests greater than 2 times normal)
* Patients on below medications due to potential interactions
* Cholesterol medications Atorvastatin (Lipitor), Rosuvastatin (Crestor), Simvastatin (Zocor), Gemfibrozil (Lopid), Niacin (Niacor), etc.
* Aspirin greater than 81 mg. Taking medicines that may increase the risk of bleeding such as Coumadin (warfarin), Plavix (clopidogrel), Xarelto (rivaroxaban), Pradaxa (dabigatran), Eliquis (apixaban) or Heparin (blood thinning medications) due to their potential interaction with resveratrol
* Chronic (daily) use of non-steroidal anti-inflammatory agents (NSAIDs) such as Motrin (Ibuprofen), Advil (Ibuprofen) or Naprosyn (Naproxen) due to potential interaction with resveratrol. (Occasional use is ok). Anti-diabetic medications: Insulin, Metformin (Glucophage, Avandamet, Glibomet, etc), Rosiglitazone (Avandia), Exenatide (Byetta), Sitagliptin (Januvia), etc. Anti-hypertensive medications Metoprolol (Lopressor), Carvedilol (Coreg), Nifedipine (Procardia, Adalat), Verapamil (Verelan,Calan, Covera), Lisinopril (Prinivil, Zestril), Captopril (Capoten), Losartan (Cozaar), Irbesartan (Avapro), etc. Testosterone and estrogen supplement. Current glucocorticoid use, or up to 3 months ago (nasal, topical, ophthalmic, and inhaled use are not exclusionary)
* Participants with other major uncontrolled medical problems or, at the discretion of the PI, Participants on other long term prescription medications for chronic illness
* At the discretion of the investigators if considered unfit for the study based on medical or psycho-social conditions
* Non-English speaking participants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
IGF2 assessment by Elisa assays | Week 0, 2, 4 6
  To determine changes in the levels of IGF-II (mIGF2 or Pro-IGF2)

SECONDARY OUTCOMES:
IGFBP-3 assessment by Elisa assays | Week 0, 2, 4, 6
  To determine changes in the levels of IGFBP-3 levels

CONTACTS AND LOCATIONS:
Overall Officials: Gayathri Nagaraj, MD, Principal Investigator — Loma Linda University Cancer Center
Locations (1):
- Loma Linda University Cancer Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No